CLINICAL TRIAL: NCT04495413
Title: Assessment of the Effect of Age on Duration of Analgesia From Single-shot Femoral Nerve Blocks
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Vanessa Loland, Professor, School of Medicine, University of Washington
Other Study IDs: STUDY00008754
Record Dates: First submitted 2020-07-27; First posted 2020-07-31 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cohort study to examine the effect of age on duration of analgesia in patients receiving single-shot femoral nerve block prior to surgery, by postoperative phone follow-up questionnaire.

DETAILED DESCRIPTION:
The purpose of this study is to find out how differences in age can affect the duration of pain relief from a femoral nerve block. Complete recovery after leg surgery involves healing of tissues at the surgical site, recovery of muscle strength and range-of-motion. Some pain is normally experienced after leg surgery. At the hospital, pain is usually treated with pain medicines, and/or a nerve block procedure. A nerve block involves injecting a local anesthetic beside the nerves to numb the nerves that supply feeling to the knee joint and surrounding tissues. The choice as to whether a participant has a nerve block or not is made by the participant and their surgeon and is not determined by this research study. The study aim is to find out how long a nerve block can relieve postsurgical pain, and whether that duration is affected by the age of the participant.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age >18 years)
* American Society of Anesthesiology physical status 1-3
* Having ambulatory surgery, who have received a single-shot femoral nerve block
* Able to read and understand English
* Have access to a phone after surgery

Exclusion Criteria:

* Pediatric patients (age <18 years)
* American Society of Anesthesiology physical status >3
* Unable to read and understand English
* Unable to have access to a phone after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult ambulatory surgery patients receiving a single-shot peripheral femoral nerve block preoperatively as part of their clinical anesthesia care on day-of-surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Duration of analgesia | From time of block placement to patient to the reported end of analgesic effect, up to 72 hours
  Total duration of analgesia from peripheral femoral nerve block

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa J Loland, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center, Seattle, Washington, United States